CLINICAL TRIAL: NCT06152276
Title: SafeHeal Diverting Ileostomy Pivotal Study (SH-SOC23)
Brief Title: SafeHeal Diverting Ileostomy Pivotal Study
Acronym: SH-SOC23
Status: Active, not recruiting | Type: Observational
Sponsor: SafeHeal Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: SH-SOC23
Record Dates: First submitted 2023-11-07; First posted 2023-11-30 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2025-05

CONDITIONS: Colorectal Cancer; Stoma Ileostomy
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Standard of Care Arm: Diverting loop ileostomy following low anterior resection of colorectal cancer
  Interventions: Other: Diverting loop ileostomy

INTERVENTIONS:
Other: Diverting loop ileostomy — Diverting loop ileostomy following low anterior resection of colorectal cancer

SUMMARY:
This SafeHeal study is designed to assess the overall safety of the low anterior resection (LAR) standard of care cancer treatment by establishing a definition of major complications. The current literature on standard of care reports adverse events/complications but does not provide a single endpoint that can be used to compare the safety of LAR cancer treatment to alternative therapies or treatments. This study will allow for the establishment of a new single safety endpoint for LAR standard of care cancer treatment.

DETAILED DESCRIPTION:
This SafeHeal study is designed to assess the overall safety of the low anterior resection (LAR) standard of care cancer treatment by establishing a definition of major complications. The current literature on standard of care reports adverse events/complications but does not provide a single endpoint that can be used to compare the safety of LAR cancer treatment to alternative therapies or treatments. This study will allow for the establishment of a new single safety endpoint for LAR standard of care cancer treatment.

The data from this study could serve as the historical control arm data of a SafeHeal Colovac Colorectal Anastomosis Protection Device Evaluation (SAFE-3) Pivotal Study designed as a prospective, non-randomized, sequential, controlled, multicenter trial comparing the investigational device, the next generation Colovac Anastomosis Protection Device, to the standard of care (SOC), diverting ostomy.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients (18 years of age or older)
2. Eligible to undergo open or minimally invasive sphincter-sparing low anterior resection with planned diverting loop ileostomy for malignancy, based on multidisciplinary team recommendations.
3. Eastern Cooperative Oncology Group (ECOG) Performance Status ≤ 2
4. Willingness to comply with protocol-specific treatment and study visits and to sign a written Informed Consent Form

Exclusion Criteria:

Preoperative

1. History of left colitis
2. Known allergy to nickel or other components of the Colovac System (not applicable for control cohort)
3. Pregnant or nursing female subject
4. Concomitant major surgical procedure in combination with Colorectal resection (i.e., hepatectomy)
5. Any serious or uncontrolled medical disorder that, in the opinion of the investigator, may increase the risk associated with study participation, impair the ability of the participant to undergo protocol described procedures or interfere with the interpretation of study results including, but not limited to:

   1. Stage IV colorectal cancer unless curative intent R0 resection is planned AND there is no associated peritoneal disease
   2. Immunodeficiency (CD4+ count < 500 CU MM)
   3. Systemic steroid therapy within the past 6 months
   4. Systemic infection at the time of surgery or requiring systemic antimicrobial therapy up to 1 week before surgery
   5. Major surgical or interventional procedures within 30 days prior to this study or planned surgical or interventional procedures within 30 days of entry into this study
   6. Diagnosis of bowel obstruction, bowel strangulation, peritonitis, bowel perforation, intraabdominal infection, ischemic bowel, or carcinomatosis
   7. Fecal incontinence, involvement of sphincter by the neoplastic disease or evidence of extensive local disease in the pelvis seen on pre-operative imaging
   8. Severe malnutrition defined as 10% weight loss within 3 months prior to enrollment.
6. The subject is currently participating in another investigational drug or device study

   Intraoperatively:
7. Occurrence of any of the following during the colorectal surgery:

   1. Blood loss (>750 cc)
   2. Blood transfusion
   3. Any new sign of bowel ischemia
   4. Positive air leak test
   5. Inadequate bowel preparation
   6. Anastomosis location greater than 10 cm from the anal verge
   7. Any other surgical complications or intra-operative risks that may place the patient at greater risk from study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with colorectal cancer undergoing low anterior resection following by a diverting loop ileostomy.
Sampling Method: Non-Probability Sample
Enrollment: 132 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Early anastomotic complications | 9 months
  Early anastomotic complications
Overall major complications | 9 months
  Major complications

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - UMass Memorial Medical Center, Worcester, Massachusetts
  - Maimonides Medical Center, Brooklyn, New York
  - Lenox Hill Hospital, New York, New York

IPD SHARING:
Plan to Share IPD: No
Deidentified study outcomes